CLINICAL TRIAL: NCT01731847
Title: Combined Neuromuscular Electrical Stimulation (NMES) With Fiberoptic Endoscopic Evaluation of Swallowing (FEES) and Traditional Swallowing Rehabilitation in the Treatment of Stroke-related Dysphagia
Brief Title: Combined NMES,FEES and Traditional Swallowing Rehabilitation in the Treatment of Stroke-related Dysphagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Shu-Fen Sun, MD,Department of Physical Medicine and Rehabilitation, Kaohsiung Veterans General Hospital, Taiwan, Kaohsiung Veterans General Hospital.
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: VGHKS96-079
Record Dates: First submitted 2012-11-13; First posted 2012-11-22 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-11

CONDITIONS: Stroke
Keywords: dysphagia,endoscopy, electrical stimulation,stroke
MeSH Terms: conditions — Stroke; Deglutition Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- The combination group (Experimental): Patients received 12 sessions of NMES for 1 hour /day, 5 days/week within a period of 2-3 weeks. FEES was done before and after NMES for evaluation and guiding therapy. All patients subsequently received 12 sessions of traditional swallowing rehabilitation (50 minutes/day, 3 days/week) for 4 weeks.
  Interventions: Procedure: the combination group

INTERVENTIONS:
Procedure: the combination group — Patients received 12 sessions of NMES for 1 hour /day, 5 days/week within a period of 2-3 weeks. FEES was done before and after NMES for evaluation and guiding therapy. All patients subsequently received 12 sessions of traditional swallowing rehabilitation (50 minutes/day, 3 days/week) for 4 weeks.

SUMMARY:
The investigators aimed to evaluate effects of combined NMES, FEES and traditional swallowing rehabilitation in stroke patients with moderate-to-severe dysphagia.

DETAILED DESCRIPTION:
Neuromuscular electrical stimulation (NMES)and Fiberoptic endoscopic evaluation of swallowing (FEES) are both promising approaches to enhance swallowing recovery for dysphagic patients. However, there is no literature on the effectiveness of combined application of these modalities in the treatment of patients with poststroke dysphagia. The purpose of this study was to prospectively investigate whether combined NMES, FEES and traditional swallowing rehabilitation can improve swallowing functions in patients with moderate-to-severe dysphagia after stroke.

ELIGIBILITY:
Inclusion Criteria:

* age between 20-85 years old
* first-time stroke confirmed by computed tomography or magnetic resonance image
* dysphagia > 3 weeks, with preservation of the swallowing reflex
* currently on a restricted diet, with a Functional Oral Intake Scale (FOIS) score of 5 or less
* Mini-Mental State Examination (MMSE)> 21
* no obvious mental depression, receptive aphasia or cognitive impairment

Exclusion Criteria:

* progressive cerebrovascular disease or other neurologic diseases
* unstable cardiopulmonary status, serious psychologic disorder or epilepsy;
* tumors, extensive surgery or radiotherapy of the head and neck region
* cardiac pacemakers
* swallowing therapy within 2 months before participation

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-02; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Functional Oral Intake Scale (FOIS) | at 6-month follow-up
  The FOIS is a 7-point ordinal scale reflecting the dietary intake of patients with dysphagia. It has adequate reliability and validity and has been used extensively in clinical studies of dysphagia to measure functional oral intake

SECONDARY OUTCOMES:
The degree of dysphagia | at 6-month follow-up
  The degree of dysphagia was classified from grade 1 to 4 after detailed clinical swallowing evaluation including cranial nerve assessment, observations of swallowing and related movements and swallowing trials using various volumes and consistencies of food
swallowing VAS | at 6-month follow-up
  Each patient completed a perceptual evaluation of his swallowing ability using a 10-cm visual analog scale (VAS). It was rated by answering a single question: ''How do you qualify your swallowing ability?'' Scores can vary from 0 (no difficulty at all) to 10 (unable to swallow).

OTHER OUTCOMES:
global satisfaction to the combination therapy | at 6-month follow-up
  Patients were asked to rate the level of global satisfaction to the combination therapy. The rating was based on a 7-point categorical scale weighted from completely satisfied, satisfied, somewhat satisfied, no change, somewhat unsatisfied, unsatisfied to completely unsatisfied.
The occurrence of adverse events or pneumonia | at 6-month follow-up
  The occurrence of adverse events or pneumonia was recorded during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Fen Sun, MD, Principal Investigator — Department of Physical Medicine and Rehabilitation, Kaohsiung Veterans General Hospital, Taiwan; National Yang-Ming University School of Medicine, Taiwan; Chien-Wei Hsu, MD, Principal Investigator — National Yang-Ming University School of Medicine, Taiwan; Department of Internal Medicine; Kaohsiung Veterans General Hospital, Taiwan; Huey-Shyan Lin, PHD, Principal Investigator — School of Nursing, Fooyin University, Taiwan
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Mann G, Hankey GJ, Cameron D. Swallowing disorders following acute stroke: prevalence and diagnostic accuracy. Cerebrovasc Dis. 2000 Sep-Oct;10(5):380-6. doi: 10.1159/000016094. PMID 10971024
- [Background] Langmore SE, Miller RM. Behavioral treatment for adults with oropharyngeal dysphagia. Arch Phys Med Rehabil. 1994 Oct;75(10):1154-60. doi: 10.1016/0003-9993(94)90094-9. PMID 7944924
- [Background] Freed ML, Freed L, Chatburn RL, Christian M. Electrical stimulation for swallowing disorders caused by stroke. Respir Care. 2001 May;46(5):466-74. PMID 11309186
- [Background] Bulow M, Speyer R, Baijens L, Woisard V, Ekberg O. Neuromuscular electrical stimulation (NMES) in stroke patients with oral and pharyngeal dysfunction. Dysphagia. 2008 Sep;23(3):302-9. doi: 10.1007/s00455-007-9145-9. Epub 2008 Apr 25. PMID 18437464
- [Background] Leder SB. Serial fiberoptic endoscopic swallowing evaluations in the management of patients with dysphagia. Arch Phys Med Rehabil. 1998 Oct;79(10):1264-9. doi: 10.1016/s0003-9993(98)90273-8. PMID 9779682
- [Background] Crary MA, Mann GD, Groher ME. Initial psychometric assessment of a functional oral intake scale for dysphagia in stroke patients. Arch Phys Med Rehabil. 2005 Aug;86(8):1516-20. doi: 10.1016/j.apmr.2004.11.049. PMID 16084801
- [Background] Shaw GY, Sechtem PR, Searl J, Keller K, Rawi TA, Dowdy E. Transcutaneous neuromuscular electrical stimulation (VitalStim) curative therapy for severe dysphagia: myth or reality? Ann Otol Rhinol Laryngol. 2007 Jan;116(1):36-44. doi: 10.1177/000348940711600107. PMID 17305276
- [Derived] Sun SF, Hsu CW, Lin HS, Sun HP, Chang PH, Hsieh WL, Wang JL. Combined neuromuscular electrical stimulation (NMES) with fiberoptic endoscopic evaluation of swallowing (FEES) and traditional swallowing rehabilitation in the treatment of stroke-related dysphagia. Dysphagia. 2013 Dec;28(4):557-66. doi: 10.1007/s00455-013-9466-9. Epub 2013 Apr 13. PMID 23584790